CLINICAL TRIAL: NCT06217692
Title: The Effect of Nutrition Education Given to Haemodialysis Patients on Food Consumption and Diet Attitude: A Randomised Controlled Study
Brief Title: The Effect of Nutrition Education Hemodialysis Patients
Acronym: Hemodialysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bayburt University (Other)
Responsible Party: Principal Investigator, Zahide Akeren, Director, Bayburt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Researcher; Researcher (Other: BayburtU)
Record Dates: First submitted 2023-12-22; First posted 2024-01-22 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Haemodialysis Patients
MeSH Terms: interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): experimental group
  Interventions: Other: nutrition education
- control group (No Intervention): control group

INTERVENTIONS:
Other: nutrition education — nutrition education
  Arms: experimental group

SUMMARY:
type of study: Clinical trial Purpose of the study: The aim of this study was to investigate the effect of nutrition education on dietary attitudes and daily consumption of essential nutrients in patients receiving haemodialysis treatment.

DETAILED DESCRIPTION:
Patients who agree to participate in the study will be included in the experimental group and control group as a result of statistical analysis and the number of patients will be determined. Then, the patients will be assigned to the groups with the randomisation method of;simple and stratified sampling;. The experimental and control groups within the scope of the research will be determined by simple randomisation method (coin toss). In the first interview, the individuals in the training group will be administered the Individual Information Form; and the;Attitude Scale of Hemodialysis Patients towards Diet Therapy as a pre-test by the researcher using the face-to-face interview method. Then, 24-Hour Food Consumption Record will be given and all food/liquids eaten and drunk for 24 hours retrospectively will be asked to be written on this form. At this stage, the researchers will help the participants to fill in the food consumption record if needed. This process will take approximately 20 minutes and the food consumption record will be collected again. Then, the individuals in the training group will be informed about nutrition education and the first nutrition education will be started. The training will last for 4 weeks, twice a week, and the length of the training will be forty minutes. After the last of the trainings, which will last 8 times in total, the Attitude Scale of Hemodialysis Patients towards Diet Therapy will be applied as a post-test using the face-to-face interview method. In the same way, 24-Hour Food Consumption Record will be given and all food/liquids eaten and drunk for 24 hours retrospectively will be asked to be written on this form. In the control group, pretest data forms (Individual Information Form and Attitude Scale towards Diet Therapy of Haemodialysis Patients) and three-day 24-Hour Food Consumption Record will be filled out, and the Attitude Scale and three-day 24-Hour Food Consumption Record will be filled out one month later as the posttest.

ELIGIBILITY:
Inclusion Criteria:

* - Receiving treatment in the haemodialysis unit of Bayburt State Hospital, having contact addresses in electronic media,
* Maintaining haemodialysis treatment for the last 3 months
* No significant psycho-emotional problems,
* It will consist of patients who are not taking any psychotropic medication and who volunteer to participate in the study.

Exclusion Criteria:

* - Reluctance to continue co-operation,
* Moving from the haemodialysis centre to other centres for any reason,
* The emergence of acute and malignant disease,
* The need for transplantation for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-02-02 (Estimated); Study Completion 2024-08-02 (Estimated)

PRIMARY OUTCOMES:
the effect of nutrition education on dietary behaviour. | 4 mounths.
  the effect of nutrition education on dietary behaviour-Attitude Scale Towards Diet Treatment of Hemodialysis Patients
Attitude Scale Towards Diet Treatment of Hemodialysis Patients. | 4 mounths.
  Attitude Scale Towards Diet Treatment of Hemodialysis Patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Bayburt University, Bayburt, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No